CLINICAL TRIAL: NCT06420583
Title: Post Operative Pain and Oral Health Related Quality of Life Following Pulpotomy VS Extraction for the Management of Permanent First Molar With Poor Prognosis: A Randomized Clinical Trial
Brief Title: Post Operative Pain and Oral Health Related Quality of Life Following Pulpotomy VS Extraction of Permanent First Molar
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aya Amr Abo ElMagd, principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2111991
Record Dates: First submitted 2024-05-10; First posted 2024-05-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Irreversible Pulpitis
Keywords: first permanent molar; pulpotomy; extraction; oral health related quality of life; post operative pain; visual analog scale
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulpotomy (Experimental): MTA Pulpotomy
  Interventions: Procedure: MTA pulpotomy
- Extraction (Active Comparator): Extraction
  Interventions: Procedure: Extraction

INTERVENTIONS:
Procedure: MTA pulpotomy — 1. Application of rubber dam for isolation, then a standardized access cavity procedure will be performed using a large sterile round end bur in a high-speed handpiece with copious irrigation, a sharp spoon excavator will remove pulpal tissues to the orifice level, bleeding control in the pulp chamber will be achieved by using 5% sodium hypochlorite.
  2. gentle condensation of MTA mix in the pulp chamber will be done by a wet sterile cotton pellet and then the rest of the pulp chamber will be filled with Glass Ionomer restoration.
  3. The tooth will be restored with a stainless steel crown.
  Other Names: vital pulp therapy
  Arms: Pulpotomy
Procedure: Extraction — After complete Anesthetic application in the affected area, non-surgical extraction will be done.
  Arms: Extraction

SUMMARY:
The goal of this clinical trial is to compare between post operative pain and oral health related quality of life in participants receiving two treatments for first permanent mandibular molars with poor prognosis.

Group I (Experimental group): Complete Pulpotomy with the use of MTA followed by stainless steel crown.

Group II (Control group): Non-surgical extraction.

DETAILED DESCRIPTION:
The principal investigator will carry out all treatment procedures, and the patients will be assigned.

For both interventions:

1. Informed consent from participating parents.
2. Baseline records photographs, percussion test, periapical and panoramic radiographs, and personal data collection.
3. A diagnostic chart with personal, medical, and dental history will be filled
4. Baseline Oral Health related quality of life questionnaire for each participant.
5. A clinical examination will be performed to assess the clinical inclusion criteria. (Pulpal and periapical diagnoses are established after clinical examination).
6. Preoperative and Postoperative photographs will be taken.
7. The radiographic examination will be performed by taking a periapical radiograph and a Panoramic radiograph through a machine to assess the inclusion criteria. The preoperative radiograph will serve as a reference for the follow-up radiographs. Standardization of the technique to avoid any distortion in the vertical dimension and to provide reproducible images using an X-ray holding device.
8. Preoperative and postoperative radiographs in the pulp therapy group will be taken by a parallel technique using an XCP film holder (Super Bite, Hawe Neos DentalSA, Switzerland).
9. Participants will then be allocated into either one of the groups according to the indicated intervention needed as follows:
10. Administration of inferior alveolar nerve block and long buccal infiltration: Septocaine® and epinephrine 1:100,000 (Articaine HCl. 4% and Epinephrine 1:100,000 Injection) at the side of the affected tooth.

ELIGIBILITY:
Inclusion Criteria:

Children aged between 8 years and 9.5 years.

* Decayed Mandibular Permanent first molars.
* Symptomatic Mandibular permanent first molar (caries-related pulpal symptoms or hypersensitivity relating to enamel hypo mineralization)

Exclusion Criteria:

* Children who are not apparently healthy.
* Lack of informed consent by the child patient's parent.
* Patients who are allergic to any of the materials used in the procedure.
* Unable to attend follow-up visits.
* Refusal of participation.

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 42 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Post operative pain | 24 hours post operatively
  will be measured using visual analog scale (VAS) The findings suggested that 100-mm VAS ratings of 0 to 4 mm can be considered no pain; 5 to 44 mm, mild pain; 45 to 74 mm, moderate pain; and 75 to 100 mm, severe pain.

SECONDARY OUTCOMES:
Oral health related quality of life | 12 months
  will be measured using Child Oral Impact on Daily Performances. It consists of 25 items distributed among 4 domains: oral symptoms, functional limitations, emotional well-being, and social well-being. It is self-reported by 8-10-year-old children using a 5-point Likert scale, and responses range from 0-4 for each item. Total scores range from 0 to100, and higher scores indicate poorer OHRQoL

OTHER OUTCOMES:
Clinical and radiographic success | 12 months
  clinical absence of signs and symptoms of infection, inflammation, swelling , pain and mobility Radiographic absence of periapical radiolucency

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt